CLINICAL TRIAL: NCT01653392
Title: BioThrax® (Anthrax) Vaccine in Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: EBS.AVA.010 / NHRC.2012.0003
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Complications; Pregnancy Outcome; Congenital Abnormalities
Keywords: Maternal Mortality; Obstetric Labor, Premature; Eclampsia; Pre-Eclampsia; Abortion, Spontaneous; Diabetes, Gestational; Pregnancy, Ectopic; Hydatidiform Mole; Fetal death; Live birth; Still birth; Premature Birth; Sex ratio; Birth weight
MeSH Terms: conditions — Pregnancy Complications; Congenital Abnormalities; Maternal Death; Obstetric Labor, Premature; Eclampsia; Pre-Eclampsia; Abortion, Spontaneous; Diabetes, Gestational; Pregnancy, Ectopic; Hydatidiform Mole; Fetal Death; Stillbirth; Premature Birth; Birth Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anthrax Vaccine Adsorbed: Active duty women who received one or more doses of BioThrax while pregnant, with the onset of pregnancy defined as the first day of the last menstrual period, and all live born infants born to women who join the registry.
  Interventions: Biological: Observational Intervention

INTERVENTIONS:
Biological: Observational Intervention — This is an observational study, therefore no interventions are specified.

SUMMARY:
The purpose of this study is to determine if inadvertent receipt of the BioThrax vaccine during pregnancy is independently associated with adverse maternal, pregnancy, or infant health outcomes.

DETAILED DESCRIPTION:
This study will use a convenience sample and passive referral to enroll participants.

For the maternal outcome portion of the study, pregnant active duty women who consent to join the registry are expected to complete several surveys over the course of their pregnancy, including an initial enrollment survey, a follow-up survey at or after the 20th week of pregnancy, and a post-delivery survey at two weeks after their delivery due date (unless a pregnancy loss is reported in the 20 week survey).

Outcomes among infants born to women enrolled in the Registry whose pregnancies result in a livebirth will be assessed with a survey during the post-delivery contact, again at 4 months of age, with a final follow-up when the infant reaches one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Female active duty service member
* Received one or more dose of BioThrax while pregnant, with the onset of pregnancy defined as the first day of the last menstrual period.

Exclusion Criteria:

* Non-service member, non-active duty pregnant female.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active duty female service members who received one or more doses of BioThrax® while pregnant, with the onset of pregnancy defined as the first day of the last menstrual period (LMP) All live born infants born to women who join the registry.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy Outcomes | Up to 44 weeks
  Pregnancy outcomes measured include live birth, still birth, spontaneous abortion, elective termination, ectopic pregnancy, or molar pregnancy Note: Twin or higher order multiple pregnancies may have more than one outcome.
Maternal Outcomes | Up to 44 weeks
  Maternal outcomes measured include maternal death, pre-eclampsia/eclampsia, preterm labor, and gestational diabetes.
Infant Outcomes | Up to 1 year of age
  Infant outcomes measured include birth defects, infant sex ratios, preterm birth, and birth weight.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Wells, MD, Principal Investigator — Naval Health Research Center
Locations (1):
- Naval Health Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No